CLINICAL TRIAL: NCT00109967
Title: A Phase II Study of CCI-779 in Combination With Rituximab in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: CCI-779 and Rituximab in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00644; N038H; U10CA025224 (NIH); CDR0000425334 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Patients also receive rituximab IV on days 1, 8, 15, and 22 of course 1 and on day 1 only of courses 3, 5, 7, 9, and 11. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of course 3, patients undergo reevaluation. Patients achieving a CR or an unconfirmed CR (CRu) receive 2 additional courses of treatment for a total of 5 courses. Patients achieving a PR or stable disease continue study treatment as outlined above for up to 12 courses. Patients achieving a PR or stable disease who subsequently achieve a CR or CRu between courses 3 and 10 receive 2 additional courses of treatment.
  Interventions: Biological: rituximab; Drug: temsirolimus

INTERVENTIONS:
Biological: rituximab — 375 mg/m^2 Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: temsirolimus — 25 mg given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase II trial is studying how well giving CCI-779 together with rituximab works in treating patients with relapsed or refractory mantle cell lymphoma. Drugs used in chemotherapy, such as CCI-779, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving CCI-779 together with rituximab may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate in patients with relapsed or refractory mantle cell lymphoma treated with CCI-779 and rituximab.

II. Determine the tolerability of this regimen in these patients by assessing toxicity.

SECONDARY OBJECTIVES:

I. Determine the time to disease progression and overall survival of patients treated with this regimen.

II. Determine the duration of response in patients treated with this regimen.

OUTLINE: Patients are stratified according to prior response to rituximab (sensitive [partial response (PR) or complete response (CR) that lasted ≥ 6 months after the last treatment with rituximab alone or in combination with chemotherapy] vs refractory [stable or progressive disease OR a PR or CR that lasted < 6 months after the last treatment with rituximab alone or in combination with chemotherapy]).

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Patients also receive rituximab IV on days 1, 8, 15, and 22 of course 1 and on day 1 only of courses 3, 5, 7, 9, and 11. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of course 3, patients undergo reevaluation. Patients achieving a CR or an unconfirmed CR (CRu) receive 2 additional courses of treatment for a total of 5 courses. Patients achieving a PR or stable disease continue study treatment as outlined above for up to 12 courses. Patients achieving a PR or stable disease who subsequently achieve a CR or CRu between courses 3 and 10 receive 2 additional courses of treatment.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed* mantle cell lymphoma (MCL)

  * Relapsed, refractory, or stable disease after prior treatment
  * Tumor must be cyclin D-1 by immunohistochemistry OR 11;14 translocation by fluorescent in situ hybridization or cytogenetics
* Measurable disease, defined as ≥ 1 of the following:

  * Unidimensionally measurable lymph node or tumor mass ≥ 2 cm by CT scan or MRI
  * Splenic enlargement if spleen is palpable ≥ 3 cm below the left costal margin
  * Malignant lymphocytosis if absolute lymphocytic count ≥ 5,000 AND lymphocytes confirmed to be monoclonal by flow cytometry
* No known central nervous system involvement (e.g., parenchymal mass or leptomeningeal involvement)
* Performance status - Eastern Cooperative Oncology Group (ECOG) 0-2
* At least 3 months
* No other concurrent treatment for MCL
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Direct bilirubin < 1.5 times ULN
* Aspartate aminotransferase (AST) ≤ 3 times ULN (5 times ULN if liver involvement by MCL is present)
* Creatinine ≤ 2 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Cholesterol ≤ 350 mg/dL
* Fasting triglycerides < 400 mg/dL
* No known HIV positivity
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other active malignancy requiring treatment OR that would preclude assessment of response to study drugs
* Prior biologic response modifiers allowed
* Prior immunotherapy allowed
* Prior high-dose therapy with stem cell support (i.e., stem cell transplantation) allowed
* No concurrent prophylactic growth factor to support neutrophils
* Prior chemotherapy allowed
* No other concurrent chemotherapy
* No concurrent corticosteroids to induce an antitumor response

  * Concurrent corticosteroids (≤ 10 mg/day of prednisone or equivalent) for adrenal insufficiency or acute allergic reactions allowed
* Prior radiotherapy allowed
* No prior treatment with a mammalian target of rapamycin (mTOR) inhibitor
* No other concurrent investigational or commercial agents or therapies for MCL
* No other concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ansell, Principal Investigator — North Central Cancer Treatment Group
Locations (195):
- United States (195):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Saint Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Carle Foundation dba Carle Cancer Center, Urbana, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - McFarland Clinic, Ames, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology - Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Merit Care Clinic Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic CCOP, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Mary's Medical Center, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health Systems, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Meritcare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cole, Sharon, K. M.D. (UIA Investigator), Kenton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Bayview Oncology Associates, Oregon, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Memorial Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Cancer Center at Saint Anne Mercy Hospital, Toledo, Ohio
  - Stark, Michael, Edward. M.D. (UIA Investigator), Toledo, Ohio
  - Toledo Clinic, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Ansell SM, Tang H, Kurtin PJ, Koenig PA, Inwards DJ, Shah K, Ziesmer SC, Feldman AL, Rao R, Gupta M, Erlichman C, Witzig TE. Temsirolimus and rituximab in patients with relapsed or refractory mantle cell lymphoma: a phase 2 study. Lancet Oncol. 2011 Apr;12(4):361-8. doi: 10.1016/S1470-2045(11)70062-6. PMID 21440503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-one patients seen at 35 sites were enrolled on this trial between May 6, 2005 and March 6, 2009. Two patients canceled before receiving treatment and 69 patients were therefore included in the analysis. There were 48 patients in group 1 (rituximab-sensitive) and 21 (rituximab-refractory) in group 2.
Pre-assignment Details: The patients were stratified by their previous response to rituximab into rituximab sensitive (group 1) or rituximab refractory (group 2) groups. Rituximab refractory was defined as no response (stable disease or progression) or a response that lasted <6 months the last time the patient received rituximab alone or rituximab with chemotherapy.
Groups:
- Group I: Rituximab Sensitive; Group II: Rituximab Refractory: Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Patients also receive rituximab IV on days 1, 8, 15, and 22 of course 1 and on day 1 only of courses 3, 5, 7, 9, and 11. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of course 3, patients undergo reevaluation. Patients achieving a CR or an unconfirmed CR (CRu) receive 2 additional courses of treatment for a total of 5 courses. Patients achieving a PR or stable disease continue study treatment as outlined above for up to 12 courses. Patients achieving a PR or stable disease who subsequently achieve a CR or CRu between courses 3 and 10 receive 2 additional courses of treatment.
  rituximab: 375 mg/m^2 Given IV
  temsirolimus: 25 mg given IV
Period: Overall Study
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory
Started | 50 | 21
Completed | 30 | 15
Not Completed | 20 | 6
Not completed — Cancel Prior to Treatment | 2 | 0
Not completed — Adverse Event | 12 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Physician Decision | 1 | 3
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory | Total
Number analyzed (Participants) | 48 | 21 | 69
Age, Continuous [Median (Full Range); unit: years] | 67.5 [51 to 86] | 66 [44 to 85] | 67 [44 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 35 | 15 | 50
Region of Enrollment [Number; unit: participants]
  United States | 48 | 21 | 69

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial Responses) as Defined by the International Workshop Criteria
Description: Complete Response (CR) - Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms.
  Partial Response (PR) requires a >=50% decrease in sum of the products of the greatest dimension (SPD) of the six largest dominant nodes or nodal masses.
  Overall Response Rate (ORR) - The number of patients who achieve a CR or PR divided by the total number of evaluable patients.
  We report the Overall Response Rate here.
Time Frame: Up to 12, 28-day cycles.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory
Number analyzed (Participants) | 48 | 21
percentage of patients | 62.5 [47.4 to 76.1] | 52.4 [29.8 to 74.3]

2. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from registration to the date of progression. Patients who died without disease progression were censored at the date of their last evaluation. Patients who were still receiving treatment at the time of these analyses were censored at the date of their last evaluation. The distribution of this time-to-event end point was estimated using the Kaplan-Meier method.
Time Frame: Patients were followed up to five years after registration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory
Number analyzed (Participants) | 48 | 21
months | 10.9 [8.0 to 12.8] | 5.4 [1.8 to 9.4]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the date of documented response to the date of progression. Patients who went off treatment due to other reasons (eg, adverse reactions, refusal of further treatment) were censored at that time. The distribution of this time-to-event end point was estimated using the Kaplan-Meier method.
Time Frame: Response duration is followed up to 5 years from registration.
Population: Of the 48 Rituximab Sensitive patients, 30 patients had a response. Of the 21 Rituximab Refractory patients, 11 patients had a response. Therefore, this endpoint uses 30 patients from the Rituximab Sensitive group and 11 patients from the Rituximab Refractory group in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory
Number analyzed (Participants) | 30 | 11
months | 11.0 [7.1 to 13.2] | 6.6 [2.0 to 20.9]

4. Secondary Outcome: Toxicity
Description: As per the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 3, toxicity was defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment by the treating physician.
  In this section, we report the number of participants that experienced at least one Grade 3 or higher adverse event.
Time Frame: Assessed during treatment (up to 12, 28-day cycles)
Measure: Number; unit: patients
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory
Number analyzed (Participants) | 48 | 21
patients
  Grade 3 or Higher | 36 | 17
  Grade 4 or Higher | 7 | 2

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from registration to death resulting from any cause. The distribution of this time-to-event end point was estimated using the Kaplan-Meier method.
Time Frame: Patients were followed for survival status for up to 5 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory
Number analyzed (Participants) | 48 | 21
months | 32.6 [24.9 to 39.7] | 24.2 [5.7 to 30.0]

ADVERSE EVENTS:
Groups:
- Group I: Rituximab Sensitive; Group II: Rituximab Refractory: temsirolimus: 25 mg given IV
Arm/Group | Group I: Rituximab Sensitive | Group II: Rituximab Refractory
Serious Adverse Events (participants affected / at risk) | 16/48 | 7/21
Other Adverse Events (participants affected / at risk) | 48/48 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I: Rituximab Sensitive (N=48) | Group II: Rituximab Refractory (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (5) | 1 (1)
Platelet count decreased (Investigations) | 3 (5) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I: Rituximab Sensitive (N=48) | Group II: Rituximab Refractory (N=21)
Hemoglobin decreased (Blood and lymphatic system disorders) | 29 (143) | 16 (88)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Endocrine disorder (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (2) | 1 (9)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (3) | 0 (0)
Watering eyes (Eye disorders) | 1 (4) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal exam abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (21) | 4 (9)
Diarrhea (Gastrointestinal disorders) | 16 (51) | 6 (10)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 1 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (3) | 3 (4)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroscopy abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 19 (47) | 5 (5)
Nausea (Gastrointestinal disorders) | 11 (20) | 10 (25)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (2)
Chest pain (General disorders) | 2 (4) | 0 (0)
Chills (General disorders) | 2 (3) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 14 (50) | 5 (18)
Fatigue (General disorders) | 36 (170) | 16 (74)
Fever (General disorders) | 4 (5) | 1 (1)
Localized edema (General disorders) | 1 (8) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (4) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Nail infection (Infections and infestations) | 1 (3) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (3)
Sinusitis (Infections and infestations) | 2 (4) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (4)
Alkaline phosphatase increased (Investigations) | 7 (25) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 4 (7)
Creatinine increased (Investigations) | 6 (30) | 5 (16)
INR increased (Investigations) | 5 (19) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (2)
Leukocyte count decreased (Investigations) | 28 (174) | 16 (68)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (64) | 3 (20)
Neutrophil count decreased (Investigations) | 21 (97) | 13 (38)
Platelet count decreased (Investigations) | 34 (176) | 15 (75)
Serum cholesterol increased (Investigations) | 35 (136) | 15 (45)
Weight loss (Investigations) | 13 (27) | 7 (26)
Anorexia (Metabolism and nutrition disorders) | 13 (27) | 9 (22)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 21 (45) | 11 (38)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (12) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 8 (28) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (7) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (6) | 4 (7)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 5 (9) | 2 (5)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (6)
Serum triglycerides increased (Metabolism and nutrition disorders) | 37 (151) | 16 (63)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (19) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (14) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (6) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 5 (15) | 2 (2)
Dysgeusia (Nervous system disorders) | 12 (30) | 2 (6)
Headache (Nervous system disorders) | 6 (8) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 4 (6) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (41) | 5 (17)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (10) | 0 (0)
Confusion (Psychiatric disorders) | 1 (6) | 1 (1)
Depression (Psychiatric disorders) | 2 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (7) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 2 (9) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 3 (3)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 3 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 5 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (14) | 2 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (12)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 10 (31) | 3 (13)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (15) | 3 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 26 (88) | 12 (40)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (7) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (9) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (6) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less